CLINICAL TRIAL: NCT05438121
Title: Drug-Coated Balloon Angioplasty Facilitates Rapid Reduction in Plaque Lipid Burden in Patients with Multivessel Coronary Artery Disease: a Serial NIRS-IVUS Imaging Study
Brief Title: STabilization of Atheroma by Lipid-reducing Effect of Drug-Coated Balloon (STABLE-DCB)
Acronym: STABLE-DCB
Status: Recruiting | Type: Observational
Sponsor: Korea University Ansan Hospital (Other)
Collaborators: B. Braun Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sunwon Kim, Sunwon Kim, MD, PhD, Associate professor, Korea University Ansan Hospital
Other Study IDs: AAG-O-H-2205
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease; Atherosclerotic Plaque; De Novo Stenosis
Keywords: drug coated balloon; Near infrared spectroscopy; NIRS-IVUS; De novo coronary lesion
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with multivessel CAD undergoing DCB PCI: I. Patients with significant multi-vessel coronary artery disease will be screened.
  II. If the patient is found to have at least one lipid-rich plaque (LRP, LCBI>250) requiring revascularization (DS>70%) will undergo multi-vessel IVUS-NIRS imaging.
  III. If multi-vessel NIRS screening revealed another LRP (LCBI>250) with DS<70%, the patient will be enrolled.
  IV. The stenotic LRP lesion (DS>70%) will be subjected to DCB angioplasty while non-stenotic LRP lesion (DS<70%) will be left unintervened and treated medically.
  V. Comparative lesions:
  1. DCB-treated LRP (DS>70%, maxLCBI>250)
  2. Unintervened, medically-treated LRP (DS<70%, maxLCBI>250)
  Interventions: Device: SeQuent Please Neo

INTERVENTIONS:
Device: SeQuent Please Neo — DCB angioplasty will be performed in accordance with the recent recommendations. Specifically, aggressive lesion predilation (balloon-to-artery ratio: 0.8 to 1.2) using either a plain balloon or a scoring balloon will be performed.

SUMMARY:
This study aims to investigate whether DCB angioplasty, compared to statin-based medical treatment alone, will lead to more reduction in plaque lipid burden as assessed by near infrared spectroscopy (NIRS) at 6-9 months following the index procedure.

DETAILED DESCRIPTION:
A large lipid core is the hallmark of coronary plaques at risk of rupture and subsequent atherothrombosis. Although statin-based medical treatment is known to regress and stabilize lipid-rich coronary plaques, it takes time for such beneficial effects to appear. This study aims to investigate whether DCB angioplasty can effectively modify de novo coronary atherosclerotic plaque and lead to reduction in plaque lipid burden as assessed by near infrared spectroscopy (NIRS) at 6-9 months following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant multivessel coronary artery disease requiring revascularization
* Any De novo lesions (reference vessel diameter of 2.25mm~4.0mm) suitable for DCB angioplasty
* Lesion suitable for intravascular imagings
* Written informed consent

Exclusion Criteria:

* Hemodynamically unstable or cardiogenic shock
* Left main stenotic lesion or graft vessel lesion
* Visible angiographic thrombus, not resolved by balloon angioplasty
* Pregnancy or breastfeeding
* Comorbidities with life expectancy < 12 months
* Severe coronary calcification or tortuosity, hindering timely DCB delivery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant multi-vessel coronary artery disease requiring revascularization
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of serially-assessed lipid core burden index (LCBI) change between DCB-treated lesion vs. medically-treated lesion | 6~9 month
  ΔLCBI: NIRS-assessed changes in LCBI between baseline and follow-up.

SECONDARY OUTCOMES:
Difference of serially-assessed plaque burden change between DCB-treated lesion vs. medically-treated lesion. | 6~9 month
  ΔPlaque burden: IVUS-assessed changes in plaque burden between baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sunwon Kim, MD, PhD, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleber FX, Mathey DG, Rittger H, Scheller B; German Drug-eluting Balloon Consensus Group. How to use the drug-eluting balloon: recommendations by the German consensus group. EuroIntervention. 2011 May;7 Suppl K:K125-8. doi: 10.4244/EIJV7SKA21. No abstract available. PMID 22027722
- [Background] Her AY, Shin ES, Bang LH, Nuruddin AA, Tang Q, Hsieh IC, Hsu JC, Kiam OT, Qiu C, Qian J, Ahmad WAW, Ali RM. Drug-coated balloon treatment in coronary artery disease: Recommendations from an Asia-Pacific Consensus Group. Cardiol J. 2021;28(1):136-149. doi: 10.5603/CJ.a2019.0093. Epub 2019 Sep 30. PMID 31565793
- [Background] Yerasi C, Case BC, Forrestal BJ, Torguson R, Weintraub WS, Garcia-Garcia HM, Waksman R. Drug-Coated Balloon for De Novo Coronary Artery Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Mar 10;75(9):1061-1073. doi: 10.1016/j.jacc.2019.12.046. PMID 32138967